CLINICAL TRIAL: NCT06343038
Title: Targeted Radionuclide Therapy in Metastatic Prostate Cancer Using a New PSMA Ligand Radiolabelled With Terbium-161 (161Tb-SibuDAB) - Dose Identification/Escalation Phase Ia/b Study
Acronym: PROGNOSTICS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-01868; th23Nicolas
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Castration-resistant Prostate Cancer
Keywords: Radioligand Therapy; Phase Ia/Ib; Circulating Tumour Cells; Biomarkers Development; Voxel-based 3D Dosimetry
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: In Phase Ia:
  Radiation dosimetry driven, head-to-head in cross-over design comparison of tumour and critical organ absorbed doses after sequential non-therapeutic injections of 161Tb-SibuDAB and 177Lu-PSMA-I&T in the same mCRPC patients undergoing standard 177Lu-PSMA-I&T RLT.
  In Phase Ib:
  Clinical and radiation dosimetry-based dose escalation study, with a classical 3+3 design, to identify the optimal biologic dose (injected activity) of 161Tb-SibuDAB for safe and effective RLT.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cross-Over Group A (Active Comparator): Cross-over design (n=10, random allocation at a 1:1 ratio). Event order:
  1. Injection of 1 GBq of 161Tb-SibuDAB,
  2. 3 weeks washout period,
  3. Injection of 1GBq of 177Lu-PSMA-I&T
  Interventions: Drug: Injection, 161Tb-SibuDAB,1GBq; Drug: Injection, 177Lu-PSMA-I&T, 1GBq
- Cross-Over Group B (Active Comparator): Cross-over design (n=10, random allocation at a 1:1 ratio). Event order:
  1. Injection of 1 GBq of 177Lu-PSMA-I&T,
  2. 3 weeks washout period,
  3. Injection of 1GBq of 161Tb-SibuDAB
  Interventions: Drug: Injection, 161Tb-SibuDAB,1GBq; Drug: Injection, 177Lu-PSMA-I&T, 1GBq
- Dose Escalation Study (Experimental): Arm composed of 5 patient cohorts each with 3-patients. Treatment consists of 4 cycles of 161Tb-SibuDAB based on the available MTD and DLT findings. Safety and efficacy evaluation performed after each therapy cycle.
  Interventions: Drug: Injection, 161Tb-SibuDAB, Dose Escalation

INTERVENTIONS:
Drug: Injection, 161Tb-SibuDAB,1GBq — Intravenous injection via peripheral venous catheter of ~1GBq 161Tb-SibuDAB (~200 μg / ~125 nM) in saline
  Arms: Cross-Over Group A; Cross-Over Group B
Drug: Injection, 177Lu-PSMA-I&T, 1GBq — Intravenous injection via peripheral venous catheter of ~1GBq 161Tb-SibuDAB (~100 μg / ~65 nM) in saline
  Arms: Cross-Over Group A; Cross-Over Group B
Drug: Injection, 161Tb-SibuDAB, Dose Escalation — Intravenous injection via peripheral venous catheter of 161Tb-SibuDAB in saline. The intervention comprises 4 cycles at 6-week intervals.
  The 161Tb-SibuDAB entry activity will be calculated based on dosimetry and toxicity data from the first 3 patients in Phase Ia of the study.
  The escalated or de-escalated 161Tb-SibuDAB activity for the subsequent 3-patient cohorts will be determined based on the clinical and biochemical safety information and on organ dosimetry results of the entry/previous cohort. Up to 4 escalation or de-escalation steps will be performed.
  Arms: Dose Escalation Study

SUMMARY:
Researchers will test a new treatment for prostate cancer. This treatment uses an antibody tagged with a small amount of radioactive material. Researchers believe the new antibody might work better than those used before.

In the first part of the study researchers will compare the new treatment to the old one on prostate cancer patients using very low doses, not strong enough to treat nor to cause strong adverse reactions. Each patient will eventually receive both treatments, but one at a time.

The aim of the second part of the study is to find the best dose of the new treatment for patients. This means finding the dose that offers the most benefits with the fewest side effects.

The performance of different prostate cancer diagnostic methods is also in scope of the study.

DETAILED DESCRIPTION:
Radioligand therapy (RLT) has emerged as an effective treatment of metastatic, castration resistant prostate cancer (mCRPC) for those patients having, prostate-specific membrane antigen (PSMA)-positive disease. This led to the FDA approval of 177Lu-PSMA-617 (PluvictoTM), a PSMA ligand radiolabelled with the β--particle emitter lutetium-177(177Lu). Despite the success of this treatment modality, the therapeutic response after RLT with 177Lu-based PSMA radioligands is limited and disease relapse inevitable. In addition, approximately 1/3 of the patients does not respond to 177Lu-based RLT despite PSMA-positive mCRPC.

It has been hypothesized that the insufficient absorbed dose delivery to macroscopic tumours and, in particular, to microscopic metastases with currently used 177Lu-based PSMA radioligands is the reason for the treatment failure in these patients. SibuDAB, a novel long-circulating PSMA ligand, was successfully tested in the preclinical setting in combination with terbium-161 (161Tb) that emits not only β--particles but also conversion and Auger electrons and, hence, delivers 2-4 times higher absorbed doses to microscopic tumours than 177Lu.

The researchers, therefore, propose to enhance the efficacy of PSMA-targeting RLT by using the long-circulating ligand (SibuDAB) labelled with 161Tb. The researchers expect 161Tb-SibuDAB to exhibit increased and/or prolonged tumour uptake with a higher deposition of energy (due to short ranged Auger electrons) resulting in a high linear energy transfer (LET) and, hence, relative biological effectiveness. 161Tb-SibuDAB should not only deliver the absorbed dose to the cellular nucleus (via β-- radiation) but also to the cell membrane and organelles (through the emission of conversion and Auger electrons) which, in mathematical models, leads to a 3-4-fold increased absorbed dose to single cancer cells compared to standard RLT.

ELIGIBILITY:
Inclusion Criteria:

* Consent form signed
* Male patients with age > 18 years
* Clinical indication for RLT with 177Lu-PSMA-I&T (progressive PSMA-positive mCRPC patients after androgen receptor signalling pathway inhibitor and taxan-based chemotherapy or patient unfit for chemotherapy)
* Patients will be included in Phase Ia while being under active therapy with 177Lu-PSMA-I&T (SoC) and after they have completed the first two cycles of 177Lu-PSMA-I&T RLT
* At least 3 measurable tumours on PSMA PET/CT (>1.5 cm) with sufficiently intense PSMA uptake (SUVmax>20)
* ECOG Performance status: 0-1
* Blood parameters: a) Leucocytes ≥ 3 G/L; b) Haemoglobin ≥ 100 g/L; c) Thrombocytes ≥ 100 G/L
* Estimated glomerular filtration rate (eGFR) > 45 ml/min
* Albumin > 25 g/L
* ALT, AST, AP: ≤ 5 times upper standard value
* Bilirubin ≤ 2 times upper standard value
* For male patients who are not surgically sterilized (orchiectomy or vasectomy), appropriate contraceptive measures must be taken during RLT and until 4 months after completion of RLT. As acceptable contraceptive count sexual abstinence or double contraceptive methods: hormonal contraceptive (oral, transdermal, implants or injections) in combination with barrier methods (spiral, condom, diaphragm)

Exclusion Criteria:

* Prior PSMA-targeted RLT (except for the 2 first cycles in Part Ia)
* PSMA-negative (or PSMA-negative / FDG-positive) disease
* Known intolerance against DOTA, DOTAGA, urea-based analogues or against any of the components/formulation of 177Lu-PSMA-I&T or 161Tb-SibuDAB solutions.
* Ongoing infection at the screening visit or a serious infection in the past 4 weeks
* Administration of another investigational product in the last 60 days before Visit 1 Day 1
* Prior or planed administration of a therapeutic radiopharmaceutical during 8 half-lives of the used radio-pharmaceutical's radionuclide, also during the ongoing study
* Any extensive radiotherapy involving bone marrow over the last 3 months before inclusion to the study
* Chemotherapy in the last 4 weeks before inclusion
* Any uncontrolled significant medical, psychiatric or surgical condition (active infection, unstable angina pectoris, cardiac arrhythmia, poorly controlled hypertension, poorly controlled diabetes mellitus [HbA1c ≥ 9%], uncontrolled congestive heart disease, etc.) or laboratory findings that might jeopardize the patient's safety or that would limit compliance with the objectives and assessments of the study. Any mental conditions which prevent the patient from understanding the type, extent and possible consequences of the study and/or an uncooperative attitude from the patient.
* Current history of any malignancy other than prostate cancer within 5 years of enrolment except for fully resected non-melanoma skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Tumour absorbed dose | 3, 24, 48 and 168 hours after each injection
  Comparison of median tumour absorbed dose, in Gy, after sequential injections of non-therapeutic test activity of 161Tb-SibuDAB and 177Lu-PSMA I&T in the same patients.
  Tumour absorbed dose is obtained by SPECT/CT of head, thorax, abdomen and pelvis and represents the time integrated tumour activity (3 tumours per patient). To avoid carry-over effects, a period of at least 21 days will be allowed between the two consecutive test injections.
Phase Ib: Identification of the optimal biological dose of 161Tb-SibuDAB for mCRPC RLT | baseline and 1 week, 2 weeks and 4 weeks after each injection. Long term: 6 and 12 months after RLT
  Identification of the optimal biological dose of 161Tb-SibuDAB, in GBq, for mCRPC RLT. The optimal maximum tolerated dose / biological dose will be the highest 161Tb-SibuDAB injected activity which elicits a clinically relevant adverse event grade G3 (according to CTCAE 5.0, ranging from G1 to G5 where G1 corresponds to mild AE and and G5 corresponds to AE related death) in maximal 1 patient per cohort / 1 patient in two cohorts.

SECONDARY OUTCOMES:
Phase Ia: Estimation of critical organ median absorbed doses | 3, 24, 48 and 168 hours after each injection
  Estimation of critical organ (bone marrow, kidney, salivary gland) median absorbed doses after injection of a non-therapeutic test activity of 161Tb-SibuDAB and 177Lu-PSMA I&T in the same patients. Critical organ absorbed dose is obtained by SPECT/CT of head, thorax, abdomen and pelvis and represents the time integrated tumour activity (3 tumours per patient). Blood samples are collected at each timepoint to enable bone marrow dosimetry.
Phase Ia: Estimation of the median tumour-to-critical organ absorbed dose ratios | 3, 24, 48 and 168 hours after each injection
  Estimation of the median tumour-to-critical organ absorbed dose ratios after test activity injections of 161Tb-SibuDAB and 177Lu-PSMA-I&T in same patient. The potential therapeutic index will be calculated by take the simple ratio between the median tumour doses (Outcome 1) and the corresponding critical organ doses (Outcome 3) in each patient.
Phase Ib: Cumulative median tumour and organ absorbed doses after 4 cycles of 161Tb-SibuDAB RLT | 3, 24, 48 and 168 hours after each injection
  The median cumulative tumour absorbed dose will represent the 4-cycle summation of the median tumour absorbed dose after receiving the therapeutic injected activity of 161Tb-SibuDAB. This will be normalized to the injected activity (expressed as Gy/GBq).
Phase Ib: Estimation of the "therapy index" for 161Tb-SibuDAB RLT. | 3, 24, 48 and 168 hours after each injection
  Simple radios will be calculated between the cumulative median tumour absorbed dose and the cumulative median doses of different critical organs following completion of 161Tb-SibuDAB RLT. The "therapy index" will be identified as the lowest value for the calculated ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Alin Chirindel, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland